CLINICAL TRIAL: NCT00263315
Title: Nebulized Liposomal Amphotericin B (Ambisome) Versus Nebulized Placebo for the Prophylaxis of Invasive Pulmonary Aspergillosis in Haematological Patients With Prolonged Neutropenia. A Randomized Clinical Trial.
Brief Title: Inhalation of Liposomal Amphotericin B to Prevent Invasive Aspergillosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Gilead Sciences (Industry); Nexstar Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: METC 191.137/2000/088
Record Dates: First submitted 2005-12-07; First posted 2005-12-08 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Aspergillosis
Keywords: aspergillosis; mycosis; neutropenia; primary prevention; hematologic diseases; amphotericin B; AmBisome; liposomal amphotericin B
MeSH Terms: conditions — Aspergillosis; Mycoses; Neutropenia; Hematologic Diseases

INTERVENTIONS:
Drug: nebulised liposomal amphotericin B

SUMMARY:
A Phase II/III randomized double-blind study comparing the safety and the efficacy of a weekly administration of 25 mg nebulized AmBisome with nebulized placebo solution to prevent invasive pulmonary aspergillosis in neutropenic hemato-oncologic patients.

DETAILED DESCRIPTION:
The morbidity, mortality and costs of invasive pulmonary aspergillosis (IPA) in neutropenic patients are high. An effective intervention to prevent IPA would therefore be welcome. The incidence of IPA in neutropenic hematology patients in our institution was recently estimated to be 5-10%. Currently, only HEPA filtration is routinely used for the prevention of IPA. In 1988, Schmitt et al. showed a significant delayed mortality in rat model of IPA when rats were treated with aerosolized conventional amphotericin-B (amB) two days before infection (1). Conventional amB may interfere with surfactant function in the lungs. In contrast, liposomal amphotericin-B contains phospholipids that are structurally related to surfactant and inhibits natural surfactant function only slightly. Furthermore, in rats, mean concentrations of AmB in lungs were 3.7 times higher at day one and almost 6 times higher at day seven after a single dose treatment with aerosolized liposomal amB when compared with conventional AmB (2). Only one non-placebo controlled randomized clinical trial evaluated the prophylactic use of inhalation therapy with conventional amB for the prevention of IPA and a non-significant 43% reduction was observed (3). We postulate that the weekly inhalation of liposomal AmB in neutropenic hematology patients can prevent IPA.

In this randomised placebo controlled clinical trial we compare the safety and efficacy of the administration of nebulized liposomal AmB (2x/week) with placebo for the prevention of IPA in haematological patients with an expected duration of neutropenia of >10d. To demonstrate a reduction in incidence of invasive pulmonary aspergillosis from 7% to 1%, a total of 170 neutropenic episodes in each arm will be included (power 80%, two-tailed alfa=0.05). The primary efficacy endpoint is the cumulative percentage of patients developing a proven or probable IPA. Per protocol serum galactomannan levels are monitored 2x/week and a HR-CT of the lungs will be performed for unexplained fever (>5d) unresponsive to broad-spectrum antibiotic therapy. EORTC/MSG criteria are used for diagnosis of IPA. The primary safety endpoint is a premature discontinuation of the study drug for >1week due to intolerance.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female hospitalized patients aged > 18 yr
2. The patient has a hematologic malignancy or will receive a bone-marrow transplant
3. The patient starts with a course of chemotherapy within 4 days or is already neutropenic at admission
4. The expected duration of severe neutropenia (PMN<0.5x10*9/L) following study entry is > 10 days
5. The patient is receiving oral antibiotic prophylaxis and fluconazole
6. Written informed consent has been obtained

Exclusion Criteria:

1. The patient shows evidence of a pulmonary fungal infection or a fungal sinusitis at trial entry
2. The concomitant use of systemic anti-aspergillus treatment such as itraconazole or any intravenous formulation of amphotericin B at study entry
3. Known hypersensitivity to amphotericin B
4. Any evidence of pneumonia or pneumonitis at trial entry
5. Any impossibility to use a nebulizer properly
6. Expected survival < 3 months at entry
7. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320
Dates: Start 2000-01; Study Completion 2006-05

PRIMARY OUTCOMES:
SAFETY: Discontinuation for >1week due to intolerance
EFFICACY: Proven/probable invasive pulmonary aspergillosis

SECONDARY OUTCOMES:
SAFETY STUDY:
A probably or definitely related AE of the respiratory tract (CTC grade > 2)
Any probably or definitely related AE by type and severity (CTC grade > 2)
Requirement of pre-medication to tolerate nebulization of the study drug
Spirometric changes after inhalation
EFFICACY STUDY:
Proven, probable or possible invasive pulmonary aspergillosis
A confirmed positive serum galactomannan concentration of 0.5 ng/ml or more
The use of systemic antifungal drugs (days) during the neutropenic episodes
The number of days of fever of unknown origin during neutropenia
Mortality due to a pulmonary fungal infection

CONTACTS AND LOCATIONS:
Overall Officials: Bart JA Rijnders, MD, PhD, Principal Investigator — Erasmus Medical Center; Siem de Marie, MD, PhD, Principal Investigator — Erasmus Medical Center; Jan J Cornelissen, MD, PhD, Principal Investigator — Erasmus Medical Center; Lennert Slobbe, MD, Principal Investigator — Erasmus Medical Center; A Vulto, PhD, Principal Investigator — Erasmus Medical Center; M J Becker, PhD, Principal Investigator — Erasmus Medical Center
Locations (2):
- Netherlands (2):
  - Erasmus MC centrumlocatie, Rotterdam
  - Erasmus MC locatie Daniel den Hoed, Rotterdam

REFERENCES:
- [Background] Schmitt HJ, Bernard EM, Andrade J, Edwards F, Schmitt B, Armstrong D. MIC and fungicidal activity of terbinafine against clinical isolates of Aspergillus spp. Antimicrob Agents Chemother. 1988 May;32(5):780-1. doi: 10.1128/AAC.32.5.780. PMID 3134851
- [Background] Cicogna CE, White MH, Bernard EM, Ishimura T, Sun M, Tong WP, Armstrong D. Efficacy of prophylactic aerosol amphotericin B lipid complex in a rat model of pulmonary aspergillosis. Antimicrob Agents Chemother. 1997 Feb;41(2):259-61. doi: 10.1128/AAC.41.2.259. PMID 9021176
- [Background] Schwartz S, Behre G, Heinemann V, Wandt H, Schilling E, Arning M, Trittin A, Kern WV, Boenisch O, Bosse D, Lenz K, Ludwig WD, Hiddemann W, Siegert W, Beyer J. Aerosolized amphotericin B inhalations as prophylaxis of invasive aspergillus infections during prolonged neutropenia: results of a prospective randomized multicenter trial. Blood. 1999 Jun 1;93(11):3654-61. PMID 10339471
- See also: Erasmus Medical Center website — http://www.erasmusmc.nl